CLINICAL TRIAL: NCT04420936
Title: Pragmatic Research in Healthcare Settings to Improve Diabetes and Obesity Prevention and Care for Our Program MAINTAIN PRIME (Promoting Real (World) IMplEmentation Through Care Teams).
Brief Title: Pragmatic Research in Healthcare Settings to Improve Diabetes and Obesity Prevention and Care for Our Program
Acronym: MAINTAIN PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Margaret (Molly) B. Conroy, Professor, Internal Medicine, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00132802; 1R18DK123372-01A1 (NIH)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Diabetes; Weight Loss; Diet Habit
Keywords: diabetes; weight loss; diet
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized clinical Trial with percent weight change at 24 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle coaching (Experimental)
  Interventions: Behavioral: MAINTAIN PRIME Lifestyle Coaching
- Control tracking (Active Comparator)
  Interventions: Behavioral: Control tracking

INTERVENTIONS:
Behavioral: MAINTAIN PRIME Lifestyle Coaching — Participants will receive two years patient support consisting of supportive coaching via EHR patient portal and tracking tools with EHR. Participants will also receive primary care physician (PCP) support with real time progress reports with counseling tips via EHR prior to visits, notification of weight changes greater or equal to 10 pounds, and annual PCP feedback.
  Arms: Lifestyle coaching
Behavioral: Control tracking — Participants will receive two years of patient support consisting of prevention updates via EHR patient portal and tracking tools within the EHR. Participants in this group will not receive primary care physician (PCP) support.
  Arms: Control tracking

SUMMARY:
Many people struggle not only to lose weight through changes in diet and physical activity, but also to maintain weight loss once they have achieved it. In a previous study, our team designed and deployed a weight maintenance intervention that was delivered through the patient portal of an electronic health record (EHR) and found that patients who tracked their weight, diet, and physical activity and also received coaching had better success with maintaining recent intentional weight loss than patients who tracked but did not receive coaching. The investigators propose to repeat the intervention in a new health care system and train routine health care staff (e.g., medical assistants and nurses) to be coaches, a more sustainable model that will allow ongoing intervention delivery after the proposed study ends.

This is a pragmatic randomized clinical Trial with percent weight change at 24 months as the primary outcome. This will be a 2-arm randomized trial that compares the MAINTAIN PRIME lifestyle coaching intervention to a control tracking intervention.

DETAILED DESCRIPTION:
Obesity is a major health problem in the United States and associated with increased risk of diabetes. While many behavioral interventions have led to successful short-term weight loss, very few programs focus on weight loss maintenance after intentional loss, and fewer still are applicable to routine health care settings. There is a great need for interventions that can assist with long-term maintenance of healthy body weight and be sustainably integrated into existing health care teams. The investigators have developed and tested an innovative weight loss maintenance intervention - Maintaining Activity and Nutrition through Technology-Assisted Innovation in Primary Care (MAINTAIN-pc) - delivered through the electronic health record (EHR) to help patients maintain recent intentional weight loss and successful lifestyle strategies.

The investigators have conducted and published a randomized clinical trial of MAINTAIN-pc at the University of Pittsburgh and found that participants who received EHR tracking tools and personalized coaching had significantly lower weight regain at 24 months (primary outcome) than participants who received EHR tracking tools alone. MAINTAIN-pc leveraged commonly available health information technology (HIT) tools to track participant progress and support patients and their providers in ongoing efforts to maintain weight loss. The investigators used an EHR platform (Epic) employed by many health care systems nationwide and integrated many parts of the MAINTAIN-pc protocol (e.g., patient identification, provider updates) with routine clinic workflow.

Despite the success of MAINTAIN-pc, two key questions about the practicality and sustainability of this intervention remain unanswered: (i) whether the HIT could be adapted at other sites and (ii) whether coaching could be delivered leveraging existing staff resources rather than interventionists supported by a research grant. The investigators propose a pragmatic clinical trial to test the implementation and impact of the MAINTAIN-pc protocol in routine health care settings: MAINTAIN PRIME (Promoting Real (World) IMplEmentation). MAINTAIN PRIME will be conducted in 14 primary care practices affiliated with the University of Utah and will capitalize on further advances in HIT (e.g., dashboards to track patient populations) and team-based care models to deliver the intervention with minimal support from research staff. The investigators will measure costs to inform future sustainability, and study workflow and individual, clinical, and organizational attributes to determine facilitators and barriers to successful implementation. With assistance from an External Advisory Board, the investigators will assemble an Implementation Toolkit of HIT and clinical resources to aid further dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75
* BMI of ≥ 25 prior to this intended weight loss
* Have experienced and maintained an intentional weight loss of at least 5% of body weight in the past 24 months
* Plan to maintain a University of Utah Health relationship in one of the participating primary care practices
* Have or be willing to get an account with the Epic MyHealth patient portal embedded in the electronic health record (EHR)

Exclusion Criteria:

* Medical conditions that might cause unintended weight loss such as cancer or thyroid disease
* Provider's assessment that patient is unable to safely undertake moderately intense unsupervised physical activity (the equivalent of 30 minutes of brisk walking)
* Edematous state that interferes with bodyweight assessment (e.g., severe congestive heart failure, end-stage renal disease, or ascites)
* Bariatric surgery in the last 2 years, or planned during the next 3 years
* Current or planned pregnancy in the next 3 years
* Currently breastfeeding
* Perceived lack of basic computer or Internet skills.
* Unable to attend the orientation/baseline visit or comply with the protocol procedures
* Any other underlying reason or concomitant condition, which in the opinion of the principal investigator, could confound the results of the study or put the participant at undue risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 24 months

SECONDARY OUTCOMES:
Change in BMI percentage | 24 months
Change in physical activity as measured in daily steps | 24 months
Change in physical activity as measured in minutes | 24 months
Change in dietary habits as measured by grams of fat | 24 months
Change in dietary habits as measured in calories | 24 months
Change in dietary habits as measured by validated diet habit survey score | 24 months
Change in quality of life as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire scores | 24 months
Change in quality of function as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire scores | 24 months
Change in blood pressure | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kukhareva PV, Weir CR, Cedillo M, Taft T, Butler JM, Rudd EA, Zepeda J, Zheutlin E, Kiraly B, Flynn M, Conroy MB, Kawamoto K. Design and implementation of electronic health record-based tools to support a weight management program in primary care. JAMIA Open. 2024 May 13;7(2):ooae038. doi: 10.1093/jamiaopen/ooae038. eCollection 2024 Jul. PMID 38745592